CLINICAL TRIAL: NCT02572570
Title: Clinical Investigation of a New Bulk Fill Composite Resin in the Restoration of Posterior Teeth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Attrition rate complicated by COVID-19 led to termination.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: 3M ESPE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-3097
Record Dates: First submitted 2015-09-21; First posted 2015-10-09 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-10

CONDITIONS: Dental Restoration Failure of Marginal Integrity; Dental Caries; Unrepairable Overhanging of Dental Restorative Materials; Poor Aesthetics of Existing Restoration; Secondary Dental Caries Associated With Failed or Defective Dental Restorations; Fractured Dental Restorative Materials Without Loss of Materials; Fracture of Dental Restorative Materials With Loss of Material
Keywords: Adult dental care
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posterior Composite Resin Restoration (Experimental): Participants will receive two commercially available tooth-colored restorative materials used for direct restoration as per manufacturer's instructions.
  Interventions: Device: Filtek Bulk Fill Posterior; Device: Filtek Supreme Ultra

INTERVENTIONS:
Device: Filtek Bulk Fill Posterior — Tooth (teeth) affected by dental caries or with an existing defective filling restored using the materials listed (Filtek Bulk Fill Posterior). Procedures done using local anesthesia and following ordinary restorative techniques.
  Other Names: Dental filling
Device: Filtek Supreme Ultra — Tooth (teeth) affected by dental caries or with an existing defective filling restored using the materials listed (Filtek Supreme Ultra). Procedures done using local anesthesia and following ordinary restorative techniques.
  Other Names: Dental filling

SUMMARY:
Polymerization shrinkage remains one of the primary disadvantages of composite resin restorative materials (tooth-colored fillings). To minimize the effects of polymerization shrinkage in the restorative treatment, the 3M ESPE company has developed a composite resin called Filtek Bulk Fill Posterior Restorative. Its decreased polymerization shrinkage and properties allow the material to be inserted in one single increment, expediting treatment. This clinical trial is designed to evaluate the performance of the new bulk fill composite resin in Class II (two-surface posterior) fillings.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age and older
* Have a pair of similar cavities or failed dental fillings in vital permanent posterior teeth requiring treatment
* Be capable of giving written informed consent.

Exclusion Criteria:

* Have a self-reported history of any adverse reaction to materials of the types to be evaluated
* Have a medical or dental history that could possibly complicate the provision of the proposed treatment and/or influence the behavior and performance of the treatment in clinical service.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-12; Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rick Walter, DDS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill School of Dentistry, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Restoration
Groups:
- Posterior Composite Resin Restoration: Posterior teeth were restored with two tooth-colored restorative materials using different techniques. Increments that were either up to 2 mm or 5 mm were placed. Twenty-two participants received one restoration and five participants received two restorations of each material, for a total of 64 restorations in 27 patients.
Period: Overall Study
Arm/Group | Posterior Composite Resin Restoration
Started | 27; 64 Restoration
Filtek Bulk Fill Posterior | 27; 32 Restoration
Filtek Supreme Ultra | 27; 32 Restoration
1 Year Follow-Up | 20; 46 Restoration
2 Year Follow-Up | 13; 34 Restoration
3 Year Follow-Up | 5; 12 Restoration
5 Year Follow-Up | 0; 0 Restoration
Completed | 0; 0 Restoration
Not Completed | 27; 64 Restoration
Not completed — Study Terminated | 27

BASELINE CHARACTERISTICS:
Units Other Than Participants: Restorations
Arm/Group | Posterior Composite Resin Restoration
Number analyzed (Participants) | 27
Number analyzed (Restorations) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Restoration Percent Success at Day 1
Description: The World Dental Federation (FDI) rates 16 categories on a scale of 1 to 5 with 1 being "Clinically Excellent" and 5 being "Clinically Poor". Scores 1-3 were considered clinically acceptable while scores 4 and 5 were considered failures. Cases were considered successful if each of the 16 following FDI criteria presented an individual score of 3 or less:
  A.Esthetic Properties Surface lustre [Item 1] Surface staining [Item 2] Color stability and translucency [Item 3] Anatomic form [Item 4] B.Functional Properties Fractures and retention [Item 5] Marginal adaptation [Item 6] Wear [Item 7] Contact point/food impact [Item 8] Radiographic examination [Item 9] Patient's view [Item 10] C.Biological Properties Postoperative (hyper)sensitivity and tooth vitality [Item 11] Recurrence of caries, erosion, abfraction [Item 12] Tooth integrity [Item 13] Periodontal response [Item 14] Adjacent mucosa [Item 15] Oral and general health [Item 16]
Time Frame: Assessed immediately post restoration placement completion
Measure: Number; unit: percentage of scores =/<3
Units Other Than Participants: Restorations
Groups:
- Filtek Bulk Fill Posterior: Dental material for posterior restoration placed in increments up to 5 mm in thickness.
- Filtek Supreme Ultra: Dental material for posterior restoration placed in increments up to 2 mm in thickness.
Arm/Group | Filtek Bulk Fill Posterior | Filtek Supreme Ultra
Number analyzed (Participants) | 27 | 27
Number analyzed (Restorations) | 32 | 32
percentage of scores =/<3 | 100 | 100

2. Primary Outcome: Restoration Percent Success at Year 1
Description: The World Dental Federation (FDI) rates 16 categories on a scale of 1 to 5 with 1 being "Clinically Excellent" and 5 being "Clinically Poor". Scores 1-3 were considered clinically acceptable while scores 4 and 5 were considered failures. Cases were considered successful if each of the 16 following FDI criteria presented an individual score of 3 or less:
  A.Esthetic Properties
  * Surface lustre [Item 1]
  * Surface staining [Item 2]
  * Color stability and translucency [Item 3]
  * Anatomic form [Item 4]
  B.Functional Properties
  * Fractures and retention [Item 5]
  * Marginal adaptation [Item 6]
  * Wear [Item 7]
  * Contact point/food impact [Item 8]
  * Radiographic examination [Item 9]
  * Patient's view [Item 10]
  C.Biological Properties
  * Postoperative (hyper)sensitivity and tooth vitality [Item 11]
  * Recurrence of caries, erosion, abfraction [Item 12]
  * Tooth integrity [Item 13]
  * Periodontal response [Item 14]
  * Adjacent mucosa [Item 15]
  * Oral and general health [Item 16]
Time Frame: Year 1
Population: Esthetic and Functional Property data not collected for 1 restoration that was replaced due to sensitivity prior to assessment visit.
Measure: Number; unit: percentage of scores =/<3
Units Other Than Participants: Restorations
Arm/Group | Filtek Bulk Fill Posterior | Filtek Supreme Ultra
Number analyzed (Participants) | 20 | 20
Number analyzed (Restorations) | 23 | 23
percentage of scores =/<3
  Esthetic Properties: number analyzed (Restorations) | 22 | 23
  Esthetic Properties | 100 | 96
  Functional Properties: number analyzed (Restorations) | 22 | 23
  Functional Properties | 96 | 96
  Biological Properties | 96 | 100

3. Primary Outcome: Restoration Percent Success at Year 2
Description: The FDI rates 16 categories on a scale of 1 to 5 with 1 being "Clinically Excellent" and 5 being "Clinically Poor". Scores 1-3 were considered clinically acceptable while scores 4 and 5 were considered failures. Cases were considered successful if each of the 16 following FDI criteria presented an individual score of 3 or less:
  A.Esthetic Properties
  * Surface lustre [Item 1]
  * Surface staining [Item 2]
  * Color stability and translucency [Item 3]
  * Anatomic form [Item 4]
  B.Functional Properties
  * Fractures and retention [Item 5]
  * Marginal adaptation [Item 6]
  * Wear [Item 7]
  * Contact point/food impact [Item 8]
  * Radiographic examination [Item 9]
  * Patient's view [Item 10]
  C.Biological Properties
  * Postoperative (hyper)sensitivity and tooth vitality [Item 11]
  * Recurrence of caries, erosion, abfraction [Item 12]
  * Tooth integrity [Item 13]
  * Periodontal response [Item 14]
  * Adjacent mucosa [Item 15]
  * Oral and general health [Item 16]
Time Frame: Year 2
Population: Esthetic and Biological Property data not collected for 1 restoration due to tooth fracture resulting in full coverage restoration.
Measure: Number; unit: percentage of scores =/<3
Units Other Than Participants: Restorations
Arm/Group | Filtek Bulk Fill Posterior | Filtek Supreme Ultra
Number analyzed (Participants) | 13 | 13
Number analyzed (Restorations) | 17 | 17
percentage of scores =/<3
  Esthetic Properties: number analyzed (Restorations) | 17 | 16
  Esthetic Properties | 94 | 100
  Functional Properties | 100 | 88
  Biological Properties: number analyzed (Restorations) | 17 | 16
  Biological Properties | 100 | 100

4. Primary Outcome: Restoration Percent Success at Year 3
Description: as for outcome 3
Time Frame: Year 3
Population: Esthetic and Biological Property data not collected for 1 restoration due to tooth fracture resulting in full coverage restoration prior to Year 2 assessment.
Measure: Number; unit: percentage of scores =/<3
Units Other Than Participants: Restorations
Arm/Group | Filtek Bulk Fill Posterior | Filtek Supreme Ultra
Number analyzed (Participants) | 5 | 5
Number analyzed (Restorations) | 6 | 6
percentage of scores =/<3
  Esthetic Properties: number analyzed (Restorations) | 6 | 5
  Esthetic Properties | 67 | 100
  Functional Properties | 100 | 67
  Biological Properties: number analyzed (Restorations) | 6 | 5
  Biological Properties | 100 | 100

5. Primary Outcome: Restoration Percent Success at Year 5
Description: as for outcome 3
Time Frame: Year 5
Population: Data not collected because study was terminated.
Units Other Than Participants: Restorations
Arm/Group | Filtek Bulk Fill Posterior | Filtek Supreme Ultra
Number analyzed (Participants) | 0 | 0
Number analyzed (Restorations) | 0 | 0

ADVERSE EVENTS:
Time Frame: From time of restoration through last follow-up visit, a planned total of up to 5 years although the trial was terminated early, thus the maximum participant follow-up was through Year 3.
Groups:
- All Participants: Includes all participants, who received both interventions.
Arm/Group | Filtek Bulk Fill Posterior | Filtek Supreme Ultra | All Participants
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 3/27 | 3/27 | 3/27
Other Adverse Events (participants affected / at risk) | 7/27 | 6/27 | 7/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filtek Bulk Fill Posterior (N=27) | Filtek Supreme Ultra (N=27) | All Participants (N=27)
Rotator Cuff Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) — Surgery required
Appendicitis (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) — Surgical intervention required
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filtek Bulk Fill Posterior (N=27) | Filtek Supreme Ultra (N=27) | All Participants (N=27)
Cracked Tooth (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Tooth Sensitivity (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
Left-sided Facial Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Acid Reflux (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Tooth Pain (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Hypermobility of Joints (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT02572570/Prot_SAP_000.pdf